CLINICAL TRIAL: NCT02127853
Title: The Effect of Pretreated Gabapentin on Hyeralgesia Occurring in the Second Operation in Staged Bilateral Cataract Surgery
Brief Title: Effect of Gabapentin on Pain of the Second Cataract Surgery
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Hee-Pyoung Park, associate professor, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SerialCataractGaba
Record Dates: First submitted 2014-04-29; First posted 2014-05-01 (Estimated); Last update posted 2015-05-12 (Estimated); Status verified 2014-04

CONDITIONS: Hyperalgesia
Keywords: serial cataract surgery; hyperalgesia; gabapentin; central sensitization
MeSH Terms: conditions — Hyperalgesia | interventions — Gabapentin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Gabapentin (Experimental): gabapentin pretreatment
  Interventions: Drug: gabapentin
- Placebo (Placebo Comparator): placebo drug pretreatment
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: gabapentin — 100 mg tid of gabapentin is prescribed to the patient for 1 week after the first eye surgery
  Arms: Gabapentin
Drug: placebo — the same regimen of placebo drug is prescribed to the patient for 1 week after the first eye surgery
  Arms: Placebo

SUMMARY:
Gabapentin pretreatment may reduce hyperalgesia occurring at the second surgery in serial, bilateral cataract surgery.

DETAILED DESCRIPTION:
Hyperalgesia occurring at the second operation in bilateral eye surgery is well known, and mechanism of central sensitization might be involved. Gabapentin is known to lower the effect of central sensitization, and its effect on acute postoperative pain has been reported. Therefore, pretreatment of gabapentin after first operation may reduce the pain at second operation.

ELIGIBILITY:
Inclusion Criteria:

* Patient of ASA(American Cociety of Anesthesiology) class I, II, III between age 20 to 80, scheduled for serial bilateral cataract surgery(1 weel interval)

Exclusion Criteria:

* refuse to participate
* BMI<16 or BMI >30
* severe cardiovascular, pulmonary, renal disease
* alcohol or drug abuse
* currently taking CNS(central nervous system) inhibitory drugs
* taking antiacids
* depressive disorder pregnancy

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2014-07; Primary Completion 2016-02 (Estimated); Study Completion 2016-02 (Estimated)

PRIMARY OUTCOMES:
proportion of subjects who answer that "pain was greater" in the second eye surgery | Intra operative (pain while fluid injection to anterior chamber)

SECONDARY OUTCOMES:
perioperative pain | end of surgery, post-op 1hr at PACU, at out-patient ward, post-op 1 day
  evaluation of overall perioperative pain

OTHER OUTCOMES:
satisfaction | intra operative
  evaluation of satisfaction of both operator and patient
anxiety | baseline (at OR room arrival, just before sterile draping)
  evaluation of patient's anxiety

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Hospital, Seoul, South Korea